CLINICAL TRIAL: NCT05502874
Title: Multicenter Registry for Assessment of Markers of Early Neurological Deterioration in Primary Intracerebral Hemorrhage
Acronym: CATCH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 08268522
Record Dates: First submitted 2022-07-31; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Intracerebral Hemorrhage; Neurologic Deficits; Hemorrhagic Stroke; Hemorrhage
Keywords: Intracerebral Hemorrhage; Neurological Deterioration; Neuroimaging; Prognosis
MeSH Terms: conditions — Cerebral Hemorrhage; Neurologic Manifestations; Hemorrhagic Stroke; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter observational study will explore the risk factors of early neurological deterioration(END) in patients with primary and to investigate the association between END and outcome.

DETAILED DESCRIPTION:
Neurological deterioration affects approximately one-third of patients with primary intracerebral hemorrhage (ICH) and increases the risk of death and dependency. However, the risk factors of early neurological deterioration (END), such as biochemical parameters, neuroimaging, and systemic complications, are not well documented in primary ICH, and the effective predictors of END is unknown.

This multicenter observational study aims to seek out the risk factors of END in patients with primary ICH and to investigate the association between END and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary intracerebral hemorrhage

Exclusion Criteria:

* Patients with secondary
* Undergo surgical evacuation of hematoma；
* Presenting contraindications or refusal to MRI
* Is pregnant
* Patients refuse to be followed up for any reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with primary intrcerebral hemorrhage will be enrolled consecutively.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Early neurological deterioration (END) | 48 hours after admission
  END is defined as an increase in the total NIHSS score of ≥ 4 points within the first 48 h after admission

SECONDARY OUTCOMES:
Late neurological deterioration (LND) | 7 days
  LND is defined as an increase in the total NIHSS score of ≥ 4 points between 48h and 7 days after admission
Functional outcome | 90 days, 1 year, 2 years after admission
  Functional outcome will be assessed with modified ranking scale(mRS).Poor outcome is defined as mRS 4-6 at follow-up
Hematoma expansion | 24 hours after admission
  Hematoma volume expansion of at least 6 mL or 33% on a CT scan obtained 24 hours after admission compared with the entry scan.
The quality of life | 90 days, 1 year, 2 years after admission
  The quality of life will be assessed with the EuroQol-5D (EQ-5D) scale.
Depression status | 90 days, 1 year, 2 years after admission
  Patient Health Questionnaire (PHQ)-9 scale will be evaluated, and higher scores means a worse status.
Cognitive function | 90 days, 1 year, 2 years after admission
  Telephone Interview for Cognitive Status-Modified(TICS-m) scale will be evaluated via telephone interview.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No